CLINICAL TRIAL: NCT03811834
Title: A Phase 1 Study to Assess Absolute Bioavailability of TAK-788 and to Characterize Mass Balance, Pharmacokinetics, Metabolism, and Excretion of [14C]-TAK-788 in Male Healthy Subjects
Brief Title: A Study to Assess Absolute Bioavailability (ABA) of Mobocertinib (TAK-788) and to Characterize Mass Balance, Pharmacokinetics (PK), Metabolism, and Excretion of Carbon-14 ([14C])-Mobocertinib in Male Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TAK-788-1002; U1111-1223-7593 (Other: WHO)
Record Dates: First submitted 2019-01-18; First posted 2019-01-22 (Actual); Results first posted 2021-07-30 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — mobocertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mobocertinib 160 mg and [14C]-Mobocertinib 50 mcg + [14C]-Mobocertinib 160 mg (Experimental): Mobocertinib 160 mg, capsule, orally, once under fasted state, followed by [14C]-mobocertinib 50 mcg (approximately 2 microcurie [mcCi]), infusion, intravenously, once on Day 1 of Period 1, further followed by a washout period of 9 days, followed by [14C]-mobocertinib 160 mg (approximately 100 mcCi), solution, orally, once under fasted state on Day 1 of Period 2.
  Interventions: Drug: Mobocertinib

INTERVENTIONS:
Drug: Mobocertinib — Mobocertinib capsule, [14C]-Mobocertinib intravenous infusion, [14C]-Mobocertinib oral solution.
  Other Names: TAK-788

SUMMARY:
The purpose of this study is to determine:

Period 1 (ABA): ABA of mobocertinib following single microdose intravenous administration of 50 microgram (mcg) (approximately 2 microcurie [mcCi]) [14 C]-]-mobocertinib and single oral administration of 160 milligram (mg) mobocertinib.

Period 2 (absorption, distribution, metabolism, and elimination [ADME]): the mass balance and metabolic profile of mobocertinib in plasma, urine, and feces, to characterize the PK of mobocertinib and its metabolites (AP32960 and AP32914) in plasma, whole blood, and urine, and total radioactivity concentration equivalents in plasma and whole blood following a single oral administration of 160 mg (approximately 100 mcCi) [14C]-mobocertinib solution.

DETAILED DESCRIPTION:
The drug being tested in this study is called mobocertinib. The study will determine ABA of mobocertinib following single microdose of 50 mcg [14C]-mobocertinib and single oral administration of 160 mg mobocertinib and will assess the mass balance and metabolic profile of mobocertinib in plasma, urine, and feces following a single oral administration of 160 mg [14C]-mobocertinib solution, and will characterize the PK of mobocertinib and its metabolites in plasma, whole blood, and urine, and total radioactivity concentration equivalents in plasma and whole blood following a single dose of 160 mg [14C]-mobocertinib.

The study will enroll approximately 6 participants. The study is designed to consist of 2 periods: Period 1 (ABA study period) and Period 2 (ADME study period). In Period 1, all participants will receive single unlabeled oral 160 mg dose of mobocertinib as capsules. At 3.75 hours post oral dosing, participants will receive 15-minute intravenous infusion of a microdose of 50 mcg (approximately 2mcCi) [14C]-mobocertinib. In Period 2, participants will receive single dose of 160 mg (approximately 100 mcCi) [14C]-mobocertinib as an oral solution.

This single center trial will be conducted in the United States. The overall time to participate in this study is approximately 65 days including screening period. Participants will be contacted approximately 30 days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Continuous non smoker who has not used nicotine containing products for at least 20 years prior to the first dosing and throughout the study, based on subject self-reporting.
2. Body mass index greater than or equal to (>=)18 and less than (˂) 30.0 kilogram per square meter (kg/m^2) at screening.

Exclusion Criteria:

1. Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. Has history or presence of alcoholism or drug abuse within the past 2 years prior to the first dosing.
3. Has positive urine drug or alcohol results at screening or first check in.
4. Estimated creatinine clearance < 80 milliliter per minute (mL/min) at screening.
5. Has tattoo(s) or scarring at or near the site of intravenous (IV) infusion or any other condition which may interfere with infusion site examination, in the opinion of the investigator.
6. Has infrequent bowel movements (less than approximately once per day) within 30 days prior to first dosing.
7. Has recent history of abnormal bowel movements, such as diarrhea, loose stools, or constipation, within 2 weeks of first dosing.
8. Has received radiolabeled substances or has been exposed to radiation sources within 12 months of first dosing or is likely to receive radiation exposure or radioisotopes within 12 months of first dosing such that participation in this study would increase their total exposure beyond the recommended levels considered safe (that is., weighted annual limit recommended by the Commission on Radiological Protection [ICRP] of 3000 millirem).
9. Donation of blood or significant blood loss within 56 days prior to the first dosing.
10. Plasma donation within 7 days prior to the first dosing.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 7 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites)

REFERENCES:
- [Derived] Hanley MJ, Zhang S, Griffin R, Zhu SX, Fram RJ, Lin J, Venkatakrishnan K, Gupta N. A phase 1 study to assess the absolute bioavailability, mass balance, pharmacokinetics, metabolism, and excretion of [14C]-mobocertinib, an oral inhibitor of EGFR exon 20 insertion mutations, in healthy participants. Invest New Drugs. 2024 Aug;42(4):343-352. doi: 10.1007/s10637-024-01446-y. Epub 2024 May 24. PMID 38789848

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 22 January 2019 to 11 March 2019.
Pre-assignment Details: Healthy male participants were enrolled in this 2-period study to receive mobocertinib 160 milligram (mg), capsules followed by carbon-14 [14C]-mobocertinib 50 microgram (mcg), infusion in Period 1 (Absolute Bioavailability [ABA]) and [14C]-mobocertinib 160 mg, solution in Period 2 (Absorption, Distribution, Metabolism, and Elimination [ADME]).
Period: Period 1 ( 7 Days)
Arm/Group | Mobocertinib 160 mg and [14C]-Mobocertinib 50 mcg + [14C]-Mobocertinib 160 mg
Started | 7
Completed | 6
Not Completed | 1
Not completed — Adverse Event | 1
Period: Washout Period (9 Days)
Arm/Group | Mobocertinib 160 mg and [14C]-Mobocertinib 50 mcg + [14C]-Mobocertinib 160 mg
Started | 6
Completed | 6
Not Completed | 0
Period: Period 2 (10 Days)
Arm/Group | Mobocertinib 160 mg and [14C]-Mobocertinib 50 mcg + [14C]-Mobocertinib 160 mg
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The safety set included all participants who received at least one dose of study drug.
Groups:
- Mobocertinib 160 mg and [14C]-Mobocertinib 50 mcg +[14C]-Mobocertinib 160 mg: Mobocertinib 160 mg, capsule, orally, once under fasted state, followed by [14C]-mobocertinib 50 mcg (approximately 2 mcCi), infusion, intravenously, once on Day 1 of Period 1, further followed by a washout period of 9 days, followed by [14C]-mobocertinib 160 mg (approximately 100 mcCi), solution, orally, once under fasted state on Day 1 of Period 2.
Arm/Group | Mobocertinib 160 mg and [14C]-Mobocertinib 50 mcg +[14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (12.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7
Weight [Mean (Standard Deviation); unit: kilogram (Kg)] | 83.74 (6.141)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 175.9 (4.14)
Body mass index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 27.079 (1.6520)

OUTCOME MEASURES:

1. Primary Outcome: Period 1: Percent Absolute Oral Bioavailability (%F) for Mobocertinib
Description: Absolute bioavailability (F), defined as the fraction or percentage of the unchanged, orally administered dose that is systemically available, relative to the total dose administered intravenously. Percent Absolute Oral Bioavailability (%F) was calculated as dose of [14C]-mobocertinib intravenous in mg*AUC∞ of mobocertinib (oral)/dose of mobocertinib (oral)* AUC∞ of [14C]-mobocertinib (intravenous)*100.
Time Frame: Day 1 pre-dose and at multiple time points (up to 144 hours) post-dose
Population: The pharmacokinetic (PK) set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile. This outcome measure (OM) was planned to be assessed only in Period 1.
Measure: Geometric Mean (90% Confidence Interval); unit: percentage bioavailability
Groups:
- Mobocertinib 160 mg and [14C]-Mobocertinib 50 mcg: Mobocertinib 160 mg, capsule, orally, once under fasted state, followed by [14C]-mobocertinib 50 mcg (approximately 2 mcCi), infusion, intravenously, once on Day 1 of Period 1.
Arm/Group | Mobocertinib 160 mg and [14C]-Mobocertinib 50 mcg
Number analyzed (Participants) | 6
percentage bioavailability | 36.7 [22.4 to 60.2]

2. Primary Outcome: Period 2: Percentage of Total Radioactivity (Cum%Dose) Recovered in Urine Relative to the Administered Radioactive Dose
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: The PK set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile. This OM was planned to be assessed only in Period 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of radioactive dose
Groups:
- [14C]-Mobocertinib 160 mg: [14C]-mobocertinib 160 mg (approximately 100 mcCi), solution, orally, once under fasted state on Day 1 of Period 2.
Arm/Group | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 6
percentage of radioactive dose | 3.57 (12.6)

3. Primary Outcome: Period 2: Percentage of Total Radioactivity (Cum%Dose) Recovered in Feces Relative to the Administered Radioactive Dose
Time Frame: Day 1 pre-dose and at multiple time points (up to 432 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of radioactive dose
Arm/Group | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 6
percentage of radioactive dose | 76.0 (6.5)

4. Primary Outcome: Period 2: Amount of Total Radioactivity Excreted in Urine (Ae[UR])
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram equivalent (mg eq)
Groups:
- [14C]-Mobocertinib 160 mg: [14C]-mobocertinib160 mg (approximately 100 mcCi), solution, orally, once under fasted state on Day 1 of Period 2.
Arm/Group | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 6
milligram equivalent (mg eq) | 5.777 (12.6)

5. Primary Outcome: Period 2: Amount of Total Radioactivity Excreted in Feces (Ae[Fe])
Time Frame: Day 1 pre-dose and at multiple time points (up to 432 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg eq
Arm/Group | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 6
mg eq | 123.1 (6.1)

6. Primary Outcome: Period 2: Percentage of Administered Radioactive Dose (%Dose) Excreted in Urine for Mobocertinib
Time Frame: Day 1: Pre-dose, 0-12 hours (hrs), 12-24 hrs, 24-48 hrs, 48-72 hrs, 72-96 hrs, 96-120 hrs, 120-144 hrs, 144-168 hrs, 168-192 hrs, 192-216 hrs, 216-240 hrs post-dose
Population: The PK set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile. Here number analyzed "n" are the participants who were evaluable for the outcome measure at given timepoints. This OM was planned to be assessed only in Period 2.
Measure: Mean (Standard Deviation); unit: percentage of radioactive dose
Arm/Group | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 6
percentage of radioactive dose
  Pre-dose | 0.00 (0.00)
  0-12 hours | 1.061 (0.22924)
  12-24 hours | 0.7462 (0.15716)
  24-48 hours | 0.7364 (0.12118)
  48-72 hours | 0.3443 (0.051037)
  72-96 hours | 0.2173 (0.040842)
  96-120 hours | 0.1425 (0.027883)
  120-144 hours | 0.1050 (0.021753)
  144-168 hours | 0.07582 (0.041180)
  168-192 hours | 0.07517 (0.012835)
  192-216 hours: number analyzed (Participants) | 5
  192-216 hours | 0.05243 (0.029772)
  216-240 hours: number analyzed (Participants) | 5
  216-240 hours | 0.05137 (0.029359)

7. Primary Outcome: Period 2: Percentage of Administered Radioactive Dose (%Dose) Excreted in Feces for Mobocertinib
Time Frame: Day 1: at Pre-dose, 0-24 hours (hrs), 24-48 hrs, 48-72 hrs, 72-96 hrs, 96-120 hrs, 120-144 hrs, 144-168 hrs, 168-192 hrs, 192-216 hrs, 216-240 hrs; 240-264 hrs, 264-288 hrs, 288-312 hrs, 213-408 hrs and 408-432 hrs
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of radioactive dose
Arm/Group | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 6
percentage of radioactive dose
  Pre-dose | 0.00 (0.00)
  0-24 hours | 16.13 (16.772)
  24-48 hours | 27.78 (19.584)
  48-72 hours | 16.10 (21.089)
  72-96 hours | 4.214 (5.3488)
  96-120 hours | 3.066 (2.8311)
  120-144 hours | 1.638 (1.8080)
  144-168 hours | 2.756 (3.3943)
  168-192 hours | 0.9919 (0.83406)
  192-216 hours: number analyzed (Participants) | 5
  192-216 hours | 2.069 (1.0034)
  216-240 hours: number analyzed (Participants) | 5
  216-240 hours | 1.695 (1.1513)
  240-264 hours: number analyzed (Participants) | 2
  240-264 hours | 0.1056 (0.14927)
  264-288 hours: number analyzed (Participants) | 2
  264-288 hours | 0.2216 (0.31341)
  288-312 hours: number analyzed (Participants) | 1
  288-312 hours | 0.7632 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  312-408 hours: number analyzed (Participants) | 1
  312-408 hours | 0.3107 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  408-432 hours: number analyzed (Participants) | 1
  408-432 hours | 0.1143 (NA) — Standard deviation could not be calculated because single participant was analyzed.

8. Primary Outcome: Period 2, Cmax: Maximum Observed Plasma and Whole Blood Concentration for Mobocertinib and Its Metabolites (AP32960 and AP32914)
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 6
ng/mL
  Plasma: Mobocertinib | 51.0 (34.9)
  Plasma: AP32960 | 22.7 (19.8)
  Plasma: AP32914 | 4.28 (34.7)
  Whole Blood: Mobocertinib | 40.5 (29.1)
  Whole Blood: AP32960 | 26.7 (10.6)
  Whole Blood: AP32914 | 3.05 (28.6)

9. Primary Outcome: Period 2, Tmax: Time to Reach the Maximum Plasma and Whole Blood Concentration (Cmax) for Mobocertinib and Its Metabolites (AP32960 and AP32914)
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Groups:
- [14C]-Mobocertinib 160 mg: 14C]-mobocertinib 160 mg (approximately 100 mcCi), solution, orally, once under fasted state on Day 1 of Period 2.
Arm/Group | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 6
hours
  Plasma: Mobocertinib | 6.00 [3.00 to 6.00]
  Plasma: AP32960 | 4.00 [3.00 to 5.00]
  Plasma: AP32914 | 6.00 [3.00 to 6.00]
  Whole Blood: Mobocertinib | 5.01 [2.01 to 6.01]
  Whole Blood: AP32960 | 5.01 [3.02 to 5.01]
  Whole Blood: AP32914 | 5.01 [4.01 to 6.01]

10. Primary Outcome: Period 2: t(1/2): Terminal Disposition Phase Half-life of Mobocertinib and Its Metabolites (AP32960 and AP32914) in Plasma and Whole Blood
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 6
hours
  Plasma: Mobocertinib | 22.8 (26.6)
  Plasma: AP32960 | 30.5 (21.1)
  Plasma: AP32914 | 14.0 (30.6)
  Whole Blood: Mobocertinib | 20.5 (25.4)
  Whole Blood: AP32960 | 30.9 (12.1)
  Whole Blood: AP32914 | 12.8 (23.1)

11. Primary Outcome: Period 2, AUC∞: Area Under the Plasma and Whole Blood Concentration-time Curve From Time 0 to Infinity for Mobocertinib and Its Metabolites (AP32960 and AP32914)
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 6
nanogram*hour per milliliter (ng*hr/mL)
  Plasma: Mobocertinib | 956 (38.6)
  Plasma: AP32960 | 486 (26.7)
  Plasma: AP32914 | 73.4 (39.9)
  Whole Blood: Mobocertinib | 729 (32.8)
  Whole Blood: AP32960 | 556 (20.2)
  Whole Blood: AP32914 | 52.4 (37.3)

12. Primary Outcome: Period 2, AUClast: Area Under the Plasma and Whole Blood Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Mobocertinib and Its Metabolites (AP32960 and AP32914)
Time Frame: Day 1 pre-dose at multiple time points (up to 240 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 6
ng*hr/mL
  Plasma: Mobocertinib | 945 (39.2)
  Plasma: AP32960 | 471 (27.5)
  Plasma: AP32914 | 63.6 (45.7)
  Whole Blood: Mobocertinib | 718 (33.2)
  Whole Blood: AP32960 | 543 (20.5)
  Whole Blood: AP32914 | 45.7 (40.4)

13. Primary Outcome: Period 2, AUCt: Area Under the Plasma and Whole Blood Concentration-time Curve From Time 0 to Time t for Mobocertinib and Its Metabolites (AP32960 and AP32914)
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 6
ng*hr/mL
  Plasma: Mobocertinib | 944.9 (39.2)
  Plasma: AP32960 | 471.1 (27.5)
  Plasma: AP32914 | 63.61 (45.7)
  Whole Blood: Mobocertinib | 717.7 (33.2)
  Whole Blood: AP32960 | 542.8 (20.5)
  Whole Blood: AP32914 | 45.74 (40.4)

14. Primary Outcome: Period 2, Cmax: Maximum Observed Plasma Radioactivity Concentration Equivalents for [14C]-Mobocertinib
Time Frame: Day 1 pre-dose at multiple time points (up to 240 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram equivalent/milliliter(ng eq/mL)
Arm/Group | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 6
nanogram equivalent/milliliter(ng eq/mL) | 1250 (13.4)

15. Primary Outcome: Period 2, Cmax: Maximum Observed Whole Blood Radioactivity Concentration Equivalents for [14C]-Mobocertinib
Time Frame: Day 1 pre-dose at multiple time points (up to 240 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram equivalent/ gram (ng eq/g)
Arm/Group | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 6
nanogram equivalent/ gram (ng eq/g) | 725 (14.6)

16. Primary Outcome: Period 2, Tmax: Time to Reach the Maximum Plasma and Whole Blood Radioactivity Concentration (Cmax) Equivalents for [14C]-Mobocertinib
Time Frame: Day 1 pre-dose at multiple time points (up to 240 hours) post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 6
hours
  Plasma | 24.0 [8.02 to 36.0]
  Whole Blood | 24.0 [8.01 to 36.0]

17. Primary Outcome: Period 2, t(1/2z): Terminal Disposition Phase Half-life of Plasma and Whole Blood Radioactivity Concentration Equivalents for [14C]-Mobocertinib
Time Frame: Day 1 pre-dose at multiple time points (up to 240 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 6
hours
  Plasma | 281 (29.1)
  Whole Blood | 301 (28.1)

18. Primary Outcome: Period 2, AUC∞: Area Under the Plasma Radioactivity Concentration Equivalents-time Curve From Time 0 to Infinity for [14C]-Mobocertinib
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram equivalent*hour per milliliter
Arm/Group | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 6
nanogram equivalent*hour per milliliter | 556000 (14.9)

19. Primary Outcome: Period 2, AUC∞: Area Under the Whole Blood Radioactivity Concentration Equivalents-time Curve From Time 0 to Infinity for [14C]-Mobocertinib
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram equivalent*hour per gram
Arm/Group | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 6
nanogram equivalent*hour per gram | 325000 (21.2)

20. Primary Outcome: Period 2, AUClast: Area Under the Plasma Radioactivity Concentration Equivalents -Time Curve From Time 0 to Last Quantifiable Concentration for [14C]-Mobocertinib
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram equivalent*hour per milliliter
Arm/Group | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 6
nanogram equivalent*hour per milliliter | 230300 (15.5)

21. Primary Outcome: Period 2, AUClast: Area Under the Whole Blood Radioactivity Concentration Equivalents -Time Curve From Time 0 to Last Quantifiable Concentration for [14C]- Mobocertinib
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram equivalent*hour per gram
Arm/Group | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 6
nanogram equivalent*hour per gram | 131000 (18.5)

22. Primary Outcome: Period 2, AUCt : Area Under the Plasma Radioactivity Concentration Equivalents-time Curve From Time 0 to Time t for [14C]-Mobocertinib
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram equivalent*hour per milliliter
Groups:
- [14C]-Mobocertinib160 mg: [14C]-mobocertinib 160 mg (approximately 100 mcCi), solution, orally, once under fasted state on Day 1 of Period 2.
Arm/Group | [14C]-Mobocertinib160 mg
Number analyzed (Participants) | 6
nanogram equivalent*hour per milliliter | 145400 (35.3)

23. Primary Outcome: Period 2, AUCt : Area Under the Whole Blood Radioactivity Concentration Equivalents-time Curve From Time 0 to Time t for [14C]-Mobocertinib
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram equivalent*hour per gram
Arm/Group | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 6
nanogram equivalent*hour per gram | 70190 (32.4)

24. Primary Outcome: Period 2, Aet1-t2: Amount of Unchanged Drug Excreted in the Urine in Each Collection Interval From t1 to t2 for Mobocertinib and Its Metabolites (AP32960 and AP32914)
Time Frame: Day 1: at Pre-dose, 0-12 hours (hrs), 12-24 hrs, 24-48 hrs, 48-72 hrs, 72-96 hrs, 96-120 hrs, 120-144 hrs, 144-168 hrs, 168-192 hrs, 192-216 hrs and 216-240 hrs post dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 6
mg
  Mobocertinib: Pre-dose | 0.001072 (0.0010474)
  Mobocertinib: 0 to 12 hours | 0.1917 (0.10878)
  Mobocertinib: 12 to 24 hours | 0.2047 (0.084347)
  Mobocertinib: 24 to 48 hours | 0.1628 (0.050589)
  Mobocertinib: 48 to 72 hours | 0.05069 (0.029114)
  Mobocertinib: 72 to 96 hours | 0.02087 (0.013052)
  Mobocertinib: 96 to 120 hours | 0.01028 (0.0052244)
  Mobocertinib: 120 to 144 hours | 0.005860 (0.0055472)
  Mobocertinib: 144 to 168 hours | 0.002438 (0.0014131)
  Mobocertinib: 168 to 192 hours | 0.0009682 (0.0011637)
  Mobocertinib: 192 to 216 hours: number analyzed (Participants) | 5
  Mobocertinib: 192 to 216 hours | 0.0009890 (0.00090295)
  Mobocertinib: 216 to 240 hours: number analyzed (Participants) | 5
  Mobocertinib: 216 to 240 hours | 0.0002824 (0.00063158)
  AP32960: Pre-dose | 0.005308 (0.0045461)
  AP32960: 0-12 hours | 0.2948 (0.078117)
  AP32960: 12-24 hours | 0.2199 (0.056834)
  AP32960: 24-48 hours | 0.2166 (0.049030)
  AP32960: 48-72 hours | 0.09444 (0.020647)
  AP32960: 72-96 hours | 0.05401 (0.014311)
  AP32960: 96-120 hours | 0.03017 (0.0070669)
  AP32960: 120-144 hours | 0.01764 (0.0068670)
  AP32960: 144-168 hours | 0.01082 (0.0028229)
  AP32960: 168-192 hours | 0.007272 (0.0023649)
  AP32960: 192-216 hours: number analyzed (Participants) | 5
  AP32960: 192-216 hours | 0.005427 (0.0021935)
  AP32960: 216-240 hours: number analyzed (Participants) | 5
  AP32960: 216-240 hours | 0.004235 (0.0016891)
  AP32914: Pre-dose | 0.00 (0.00)
  AP32914: 0-12 hours | 0.08336 (0.022896)
  AP32914: 12-24 hours | 0.06029 (0.015305)
  AP32914: 24-48 hours | 0.04953 (0.021338)
  AP32914: 48-72 hours | 0.01543 (0.0068257)
  AP32914: 72-96 hours | 0.005859 (0.0040117)
  AP32914: 96-120 hours | 0.002477 (0.0016606)
  AP32914: 120-144 hours | 0.0008353 (0.0010134)
  AP32914: 144-168 hours | 0.0001780 (0.00043613)
  AP32914: 168-192 hours | 0.00 (0.00)
  AP32914: 192-216 hours: number analyzed (Participants) | 5
  AP32914: 192-216 hours | 0.00 (0.00)
  AP32914: 216-240 hours: number analyzed (Participants) | 5
  AP32914: 216-240 hours | 0.00 (0.00)

25. Primary Outcome: Period 2, CLR: Renal Clearance for Mobocertinib and Its Metabolites (AP32960 and AP32914)
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour ( L/h)
Arm/Group | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 6
liter per hour ( L/h)
  Mobocertinib | 0.657 (44.3)
  AP32960 | 1.95 (22.5)
  AP32914 | 2.85 (27.9)

26. Primary Outcome: Period 2, Percentage Change of [14C]-Radioactivity in Whole Blood Relative to Plasma Over the Time for [14C]-Mobocertinib, (Whole Blood : Plasma Partitioning Ratio)
Time Frame: At 0.5 hours (hrs), 1 hr, 2 hrs, 3 hrs, 4 hrs, 5 hrs, 6 hrs, 8 hrs, 12 hrs, 24 hrs, 36 hrs, 48 hrs, 72 hrs, 96 hrs, 120 hrs, 144 hrs, 168 hrs, 192 hrs, 216 hrs and 240 hrs post-dose
Population: The PK set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile. Here number analyzed "n" are the participants who were evaluable for the outcome measure at given timepoints. Here, '0' in the number analyzed field signifies that no participants were evaluable at specified time points. This OM was planned to be assessed only in Period 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 6
ratio
  At 0.5 hour | 1.022 (21.9)
  At 1 hour | 0.9851 (36.0)
  At 2 hours | 0.9055 (25.3)
  At 3 hours | 0.8403 (22.4)
  At 4 hours | 0.8221 (23.3)
  At 5 hours | 0.8545 (17.2)
  At 6 hours | 0.7647 (18.6)
  At 8 hours | 0.7634 (20.7)
  At 12 hours | 0.7573 (17.6)
  At 24 hours | 0.8139 (23.0)
  At 36 hours | 0.7028 (13.2)
  At 48 hours | 0.7113 (14.7)
  At 72 hours | 0.6453 (18.8)
  At 96 hours: number analyzed (Participants) | 5
  At 96 hours | 0.6164 (18.0)
  At 120 hours: number analyzed (Participants) | 4
  At 120 hours | 0.6260 (13.2)
  At 144 hours: number analyzed (Participants) | 1
  At 144 hours | 0.5946 (NA) — Geometric coefficient of variation could not be calculated because single participant was analyzed.
  At 168 hours: number analyzed (Participants) | 0
  At 192 hours: number analyzed (Participants) | 0
  At 216 hours: number analyzed (Participants) | 0
  At 240 hours: number analyzed (Participants) | 0

27. Secondary Outcome: Period 1, Ceoi: Plasma Concentration at the End of Infusion for [14C]-Mobocertinib, and Its Metabolites ([14C]-AP32960 and [14C]-AP32914)
Time Frame: Day 1 pre-dose and at multiple time points (up to 144 hours) post-dose
Population: The PK set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile. This OM was planned to be assessed only in Period 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms per milliliter (pg /mL)
Groups:
- Mobocertinib160 mg and [14C]-Mobocertinib 50 mcg: Mobocertinib 160 mg, capsule, orally, once under fasted state, followed by [14C]-mobocertinib 50 mcg (approximately 2 mcCi), infusion, intravenously over 15 minutes, once on Day 1 of Period 1.
Arm/Group | Mobocertinib160 mg and [14C]-Mobocertinib 50 mcg
Number analyzed (Participants) | 6
picograms per milliliter (pg /mL)
  [14C]-Mobocertinib | 146.3 (46.4)
  [14C]- AP32960 | 1.842 (20.5)
  [14C]- AP32914 | 2.432 (9.3)

28. Secondary Outcome: Period 1, Cmax: Maximum Observed Plasma Concentration for Mobocertinib and Its Metabolites (AP32960 and AP32914) After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 144 hours) post-dose
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Mobocertinib 160 mg and [14C]-Mobocertinib 50 mcg
Number analyzed (Participants) | 6
ng/mL
  Mobocertinib | 56.7 (52.2)
  AP32960 | 23.29 (21.2)
  AP32914 | 4.086 (36.0)

29. Secondary Outcome: Period 1, Cmax: Maximum Observed Plasma Concentration for [14C]-Mobocertinib and Its Metabolites ([14C]-AP32960 and [14C]-AP32914) After Intravenous Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 144 hours) post-dose
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Mobocertinib 160 mg and [14C]-Mobocertinib 50 mcg
Number analyzed (Participants) | 6
pg/mL
  [14C]-mobocertinib | 148 (44.0)
  [14C]-AP32960 | 6.631 (76.4)
  [14C]-AP32914 | 3.772 (33.8)

30. Secondary Outcome: Period 1, Time to Reach the Maximum Plasma Concentration (Cmax) for Mobocertinib and Its Metabolites (AP32960 and AP32914) After Oral, and [14C]-Mobocertinib and Its Metabolites ([14C]-AP32960 and [14C]-AP32914) After Intravenous Administration
Description: Data for mobocertinib and its metabolites (AP32960 and AP32914) is reported following the oral administration, and data for [14C]-mobocertinib and its metabolites ([14C]-AP32960 and [14C]-AP32914) is reported following intravenous administration.
Time Frame: Day 1 pre-dose and at multiple time points (up to 144 hours) post-dose
Population: as for outcome 27
Measure: Median (Full Range); unit: hours
Groups:
- Mobocertinib 160 mg and [14C]-Mobocertinib 50 mcg: Mobocertinib160 mg, capsule, orally, once under fasted state, followed by [14C]-mobocertinib 50 mcg (approximately 2 mcCi), infusion, intravenously, once on Day 1 of Period 1.
Arm/Group | Mobocertinib 160 mg and [14C]-Mobocertinib 50 mcg
Number analyzed (Participants) | 6
hours
  Mobocertinib | 5.00 [4.00 to 6.00]
  AP32960 | 4.502 [4.00 to 6.00]
  AP32914 | 5.000 [4.00 to 6.00]
  [14C]-mobocertinib | 0.26 [0.26 to 1.25]
  [14C]- AP32960 | 3.257 [2.25 to 8.26]
  [14C]- AP32914 | 2.26 [2.26 to 2.26]

31. Secondary Outcome: Period 1, AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Mobocertinib and Its Metabolites (AP32960 and AP32914) After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 144 hours) post-dose
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Mobocertinib 160 mg and [14C]-Mobocertinib 50 mcg
Number analyzed (Participants) | 6
ng*hr/mL
  Mobocertinib | 1050 (64.9)
  AP32960 | 478.2 (30.6)
  AP32914 | 73.02 (53.2)

32. Secondary Outcome: Period 1, AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for [14C]-Mobocertinib and Its Metabolites ( [14C]-AP32960 and [14C]-AP32914) After Intravenous Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 144 hours) post-dose
Population: The PK set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile. Here number analyzed "n" are the participants who were evaluable for the outcome measure at given timepoints. This OM was planned to be assessed only in Period 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram*hour/ milliliter (pg*hr/mL)
Arm/Group | Mobocertinib 160 mg and [14C]-Mobocertinib 50 mcg
Number analyzed (Participants) | 6
picogram*hour/ milliliter (pg*hr/mL)
  [14C]-Mobocertinib | 680 (30.4)
  [14C]- AP32960 | 187.8 (60.2)
  [14C]- AP32914: number analyzed (Participants) | 1
  [14C]- AP32914 | 89.71 (NA) — Geometric coefficient of variation could not be calculated because single participant was analyzed.

33. Secondary Outcome: Period 1, AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to Last Quantifiable Concentration for Mobocertinib and Its Metabolites (AP32960 and AP32914) After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 144 hours) post-dose
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Mobocertinib 160 mg and [14C]-Mobocertinib 50 mcg
Number analyzed (Participants) | 6
ng*hr/mL
  Mobocertinib | 1032 (65.6)
  AP32960 | 461.2 (30.1)
  AP32914 | 66.92 (53.6)

34. Secondary Outcome: Period 1, AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to Last Quantifiable Concentration for [14C]-Mobocertinib and Its Metabolites ([14C]-AP32960 and [14C]-AP32914) After Intravenous Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 144 hours) post-dose
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*hr/mL
Arm/Group | Mobocertinib 160 mg and [14C]-Mobocertinib 50 mcg
Number analyzed (Participants) | 6
pg*hr/mL
  [14C]-Mobocertinib | 617.9 (34.0)
  [14C]-AP32960 | 133.1 (63.1)
  [14C]-AP32914: number analyzed (Participants) | 2
  [14C]-AP32914 | 31.52 (113.7)

35. Secondary Outcome: Period 1, AUCt: Area Under the Plasma Concentration-time Curve From Time 0 to Time t for [14C]-Mobocertinib and Its Metabolites ([14C]-AP32960 and [14C]-AP32914) After Intravenous Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 144 hours) post-dose
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram*hour per milliliter (pg*hr/mL)
Arm/Group | Mobocertinib 160 mg and [14C]-Mobocertinib 50 mcg
Number analyzed (Participants) | 6
picogram*hour per milliliter (pg*hr/mL)
  [14C]-Mobocertinib | 617.9 (34.0)
  [14C]- AP32960 | 133.1 (63.1)
  [14C]- AP32914: number analyzed (Participants) | 2
  [14C]- AP32914 | 31.52 (113.7)

36. Secondary Outcome: Period 1, t(1/2):Terminal Disposition Phase Half-Life of Mobocertinib and Its Metabolites (AP32960 and AP32914) in Plasma After Oral, and [14C]-Mobocertinib and Its Metabolites ( [14C]-AP32960 and [14C]-AP32914) in Plasma After Intravenous Administration
Description: as for outcome 30
Time Frame: Day 1 pre-dose and at multiple time points (up to 144 hours) post-dose
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Mobocertinib 160 mg and [14C]-Mobocertinib 50 mcg
Number analyzed (Participants) | 6
hours
  Mobocertinib | 22.9 (17.9)
  AP32960 | 29.077 (18.2)
  AP32914 | 12.545 (37.5)
  [14C]-Mobocertinib | 22.2 (41.3)
  [14C]- AP32960: number analyzed (Participants) | 5
  [14C]- AP32960 | 20.317 (39.1)
  [14C]- AP32914: number analyzed (Participants) | 1
  [14C]- AP32914 | 11.900 (NA) — Geometric coefficient of variation could not be calculated because single participant was analyzed.

37. Secondary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Time Frame: Baseline up to 30 days after last dose of study drug in Period 2 (Day 41)
Population: The safety set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Mobocertinib 160 mg and [14C]-Mobocertinib 50 mcg | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 7 | 6
Participants | 6 | 4

38. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in 12-lead Electrocardiogram (ECG) Findings
Time Frame: Baseline up to 30 days after last dose of study drug in Period 2 (Day 41)
Population: The safety set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Mobocertinib 160 mg and [14C]-Mobocertinib 50 mcg | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 7 | 6
Participants | 0 | 0

39. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Time Frame: Baseline up to 30 days after last dose of study drug in Period 2 (Day 41)
Population: The safety set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Mobocertinib 160 mg and [14C]-Mobocertinib 50 mcg | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 7 | 6
Participants | 0 | 0

40. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Laboratory Values
Time Frame: Baseline up to 30 days after last dose of study drug in Period 2 (Day 41)
Population: The safety set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Mobocertinib 160 mg and [14C]-Mobocertinib 50 mcg | [14C]-Mobocertinib 160 mg
Number analyzed (Participants) | 7 | 6
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug until 30 days after last dose of study drug in Period 2 (up to Day 41)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Mobocertinib 160 mg and [14C]-Mobocertinib 50 mcg | [14C]-Mobocertinib 160 mg
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 6/7 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mobocertinib 160 mg and [14C]-Mobocertinib 50 mcg (N=7) | [14C]-Mobocertinib 160 mg (N=6)
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Eructation (Gastrointestinal disorders) | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Cow's milk intolerance (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT03811834/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT03811834/SAP_001.pdf